CLINICAL TRIAL: NCT05468203
Title: PREVENTion With Sglt-2 Inhibition of Acute Kidney Injury in Intensive Care
Acronym: PREVENTS-AKI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University Medical Center Groningen (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GI-RM-7738
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: Kidney failure; Sodium Glucose cotransporter-2 inhibitors; Critically ill; Critical Care; ICU
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency; Critical Illness | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Prospective, international, multi-centre, double blinded, randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapaliflozin 10mg tablet administered once daily while in ICU for up to 30 days
  Interventions: Drug: Dapagliflozin 10mg Tab
- Matched Placebo (Placebo Comparator): Matched placebo tablet administered once daily while in ICU for up to 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Patients will be randomly assigned to receive either dapagliflozin 10 mg or placebo daily while in ICU for up to 30 days
  Other Names: SGLT2 inhibitor
  Arms: Dapagliflozin
Drug: Placebo — Patients will be randomly assigned to receive either dapagliflozin 10 mg or placebo daily while in ICU for up to 30 days
  Arms: Matched Placebo

SUMMARY:
Background Acute Kidney Injury (AKI) is a potentially life-threatening condition caused by unsafe levels of fluid and waste products accumulating in the body. Often, patients with AKI need treatment with an artificial kidney (called renal replacement therapy or dialysis) to do the work of their kidneys and remove these dangerous levels of fluid and waste from the body. If left untreated, AKI can become a chronic (long-term) condition that may require treatment for life.

Dapagliflozin is a medication used to treat patients with diabetes, heart disease and long-term (chronic) kidney disease. Recently, Dapagliflozin has been shown to slow the progression of other kidney related complications, however this has not yet been studied in critically ill patients.

Aim To determine if giving Dapagliflozin (one tablet a day) compared to placebo (a tablet that looks identical but has no active ingredients), decreases injury to the kidneys in patients admitted to the Intensive Care Unit.

Design This study will enrol 3000 patients from 45-50 hospitals worldwide. It is a 'randomised controlled trial' meaning patients will be randomly assigned (like tossing a coin) by a computer to receive either Dapagliflozin or placebo for a maximum of 30 days whilst in the ICU. The study is also a 'double blinded trial' meaning that neither the doctor, the intensive care staff or the patient will know which study treatment they are receiving.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an increasingly common complication of hospitalisation globally, and a major driver of poor patient outcomes, including higher mortality and reduced quality of life. While numerous studies, including several led by investigators in this grant team, have tested treatments to reduce the impact of AKI, none have been shown to improve outcomes. The absence of any proven therapy highlights a critical unmet need.

A novel class of medicines, inhibitors of the sodium-glucose co-transporter II (SGLT-2 inhibitors), have been shown in recent years to have dramatic effects upon cardiovascular and renal outcomes in patients with heart failure at high risk for renal failure. The evidence suggests that these drugs might prevent AKI from occurring, but this has not been intentionally tested in adequately powered trials. A recently published randomised controlled trial evaluated the use of these drugs in acutely unwell COVID-19 patients and did not raise any safety concern in this acute setting. The trial also showed a numerically lower rate of AKI in those that received the SGLT-2 inhibitor dapagliflozin compared to placebo, but the trial was not sufficiently powered for this outcome.

The PREVENTion with Sglt2 inhibition of Acute Kidney Injury in intensive care (PREVENTS-AKI) trial, will test the effect of dapagliflozin versus placebo upon patients' risk of developing severe AKI in a population admitted to intensive care. This global trial will test the most promising treatment for mitigating the increased risk of AKI. The results will provide the first definitive insight into the prevention of AKI with these agents and will shape global clinical practice in an area where treatments are profoundly lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Admitted to ICU within the last 7 days
* Expected to be in the ICU the day after tomorrow
* An arterial or central venous catheter is in situ, or placement is planned for routine management
* Able to receive study treatment orally or via enteral route
* At least one of the following risk factors for AKI:

  * Required fluid resuscitation, defined as a bolus of fluid prescribed to be given over ≤1 hour to increase or maintain intravascular volume that is in addition to maintenance fluids
  * Being treated with continuous vasopressors or inotropes to maintain a systolic blood pressure > 90mmHg, or mean arterial blood pressure > 60mmHg or a MAP target set by the treating clinician for maintaining perfusion
* At least one of the following pre-morbid risk factors:

  * Treatment for high blood pressure
  * Treatment for type 2 diabetes (minimum diet therapy)
  * Atherosclerotic cardiovascular disease
  * History of heart failure
  * Impaired renal function, defined as an eGFR between 20 - 60 mL/min/1.73m2
  * Estimated BMI 30 kg/m2 or more
  * Age 60 years or more

Exclusion Criteria:

* Met all inclusion criteria more than 24 hours ago
* History of type 1 diabetes mellitus or diabetic ketoacidosis
* COVID-19 infection as the reason for ICU admission
* Requiring renal replacement therapy for intoxication
* eGFR less than 20 mL/min/1.73m2
* Known hypersensitivity to any SGLT-2 inhibitor e.g. dapagliflozin, canagliflozin, empagliflozin, ertugliflozin
* Solid organ transplantation within the last 12 months
* Likely to be transferred to another hospital in the next 3 days
* Known or suspected pregnancy
* Death is deemed imminent or inevitable
* Life expectancy is estimated to be less than 90 days
* Patient or the treating clinician declines to participate
* Enrolled in another interventional trial for which co-enrolment is not approved
* Patient has previously been enrolled in the PREVENTS-AKI Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: Doubling of serum creatinine from baseline, initiation of renal replacement therapy or death | Within 30 days of randomisation
  Proportion of patients experiencing a component of the composite outcome, defined as a doubling of serum creatinine from the study baseline value, initiation of RRT or death

SECONDARY OUTCOMES:
Doubling of Serum Creatinine | Within 30 days of randomisation
  Proportion of patients with a doubling of serum creatinine from baseline value
Requirement of Renal Replacement Therapy (RRT) | Within 30 days of randomisation
  Proportion of patients requiring RRT
All-cause mortality | Within 30 days of randomisation
  Proportion of patients who have died from any cause
Vasoactive drug therapy | Within 30 days of randomisation
  Proportion of patients who were treated with vasoactive drugs
Mechanical ventilation | Within 30 days of randomisation
  Proportion of patients who required mechanical ventilation
Ventricular tachycardia or ventricular fibrillation | Within 30 days of randomisation
  Proportion of patients who experienced ventricular tachycardia or ventricular fibrillation lasting at least 30 seconds whilst in intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Gallagher, MBBS, FRACP, Study Director — The George Institute
Locations (2):
- Australia (2):
  - Grampians Health, Ballarat, Victoria
  - Austin Health, Heidelberg, Victoria